CLINICAL TRIAL: NCT00572338
Title: UARK 91-004 Therapeutic Research in Multiple Myeloma
Brief Title: Therapeutic Research in Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: UARK 91-004
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * A bone marrow aspirate and biopsy
  * Blood
  * Fine Needle aspirates
  * Swabs of skin, throat, other sites
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with myeloma/related diseases
  Interventions: Other: No drugs are involved

INTERVENTIONS:
Other: No drugs are involved — No treatment or drugs are involved in this research. Participating in this study requires that blood and bone marrow samples be obtained as a part of the diagnostic work-up or follow-up of participant's multiple myeloma. Bone marrow/peripheral blood samples will be collected at the same time for research purposes. Data will be collected including demographic information gathered from your medical record, including gender, date of birth, ethnicity, date of diagnosis, laboratory and pathology results, treatment protocols, dates of relapses, subsequent treatment protocols, and current treatments and medications.
  Other Names: none, no treatment

SUMMARY:
The purpose of this study is to learn how myeloma cells grow and become a cancer, how to distinguish them from normal cells and how to eliminate these cells selectively.

DETAILED DESCRIPTION:
Participating in this study will require that blood and bone marrow samples be obtained as a part of the diagnostic work-up or follow-up of your multiple myeloma. Bone marrow/peripheral blood/tissue samples will be collected for research purposes, as well as testing for genetic traits of Castleman's disease if you consent to this study. In addition, data will be collected including demographic information gathered from your medical record, including gender, date of birth, ethnicity, date of diagnosis, laboratory and pathology results, treatment protocols, dates of relapses, subsequent treatment protocols, and current treatments and medications.

ELIGIBILITY:
Inclusion Criteria:

* Any subject evaluated for a MIRT protocol

Exclusion Criteria:

* Subjects who have not been evaluated for a MIRT protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples will be studied in the laboratory and in experimental animal models. These analyses and animal models may help to better understand multiple myeloma and to better select the appropriate treatment for all participants with multiple myeloma.
Sampling Method: Probability Sample
Enrollment: 6388 (Actual)
Dates: Start 2003-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, MD, PhD, Principal Investigator — UAMS Myeloma Institute for Research and Therapy
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States